CLINICAL TRIAL: NCT05216731
Title: Bypass Versus Endovascular Procedure in Long Lesions of the Superficial Femoral Artery in the Claudicant
Acronym: PELI-CAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP191106
Record Dates: First submitted 2022-01-24; First posted 2022-01-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lesion; Femoral
Keywords: Bypass; Endovascular procedure; Long lesions of the superficial femoral artery
MeSH Terms: interventions — Endovascular Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bypass group (Experimental): Under general or local anesthesia: Use of the best vascular substitute (inverted saphenous vein or vascular prosthesis).
  Interventions: Procedure: Femoro-popliteal bypass
- Endovascular procedure group (Active Comparator): Under general anesthesia, local anesthesia or sedation: Performing a balloon angioplasty completed by preferred stent deployment or drug-coated balloon angioplasty.
  Interventions: Procedure: Endovascular procedure

INTERVENTIONS:
Procedure: Femoro-popliteal bypass — Under general or local anesthesia: Use of the best vascular substitute (inverted saphenous vein or vascular prosthesis).
  Arms: Bypass group
Procedure: Endovascular procedure — Under general anesthesia, local anesthesia or sedation: Performing a balloon angioplasty completed by preferred stent deployment or drug-coated balloon angioplasty.
  Arms: Endovascular procedure group

SUMMARY:
In lower limb peripheral arterial disease, the stage of intermittent claudication has a prevalence of more than 5% over the age of 60, and affects patients who are often still active. Frequent anatomical lesions are strictures / occlusions of the superficial femoral artery.

There is a current low level of evidence for the treatment modalities of long lesions (15-25 cm) of the superficial femoral artery and in particular no clinical trial comparing the femoro-popliteal bypass to the endovascular procedure whose patency in retrospective series. appears lower than that of surgery but nevertheless appears in the European recommendations for first-line treatment, with the absence of a dedicated trial being highlighted.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Effective contraception for the duration of research for fertile women of childbearing age
* Unilateral Rutherford 2 or 3 symptomatic Lower Extremity Artery Disease (LEAD) arteritic patient with a lesion of the superficial femoral artery Trans-Atlantic Inter-Society Consensus (TASC) C or D between 15 and 25 cm
* Patient eligible for bypass surgery and endovascular procedure
* No alteration of the upstream flow (iliac flow preserved or restored)
* Patient with at least one patent artery below the knee
* Patient informed and having signed the information and consent form to participate in the study

Exclusion Criteria:

* Known pregnancy or breastfeeding
* Iliac flow altered upstream
* History of surgery or stent on the affected superficial femoral artery
* Concomitant bacteremia (positive blood cultures in the 7 days preceding the procedure)
* Known intolerance to antiaggregants or heparin
* Contraindication to the endovascular procedure (severe renal failure contraindicating the injection of contrast product despite prior hydration, known severe allergy to iodinated contrast product [unless the center chooses to use carbon dioxide injection]) or bypass surgery (cardiovascular, respiratory or other comorbidities, contraindicating general anesthesia, local contraindications for bypass: skin lesion at the operative site)
* No affiliation to a social security regime or to another social protection regime
* Patient deprived of liberty or under legal protection (guardianship, trusteeship)
* Inability, according to the investigator, to understand or refusal to sign the informed consent to participate in the study (non-French speaking patient, cognitive disorders)
* Ongoing participation in another research protocol Participation in non-interventional research is authorized

Secondary exclusion criterion:

* Negative opinion from the anesthesiologist-resuscitator at the end of the pre-anesthetic consultation
* Positive pregnancy test from the pre-operative laboratory test (result received after obtaining consent, but before the surgical procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2030-03-07 (Estimated); Study Completion 2030-05-20 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate at 2 year follow-up. | 2 year
  Primary patency is defined by the presence of satisfactory flow in the superior femoral artery or bypass

SECONDARY OUTCOMES:
Primary patency rate at 1 year follow-up. | 1 year
  Primary patency is defined by the presence of satisfactory flow in the superior femoral artery or bypass
Secondary patency rate at 1 and 2 years follow-up. | 1 and 2 years
  Secondary patency is defined as the patency after treatment of a (re)occlusion of the index lesion or bypass.
Clinical improvement according to the Rutherford classification (clinical stages of ischemia) at 1, 6, 12 and 24 months | 1, 6, 12 and 24 months
  Clinical improvement is considered as an improvement in the Rutherford stage, i.e. a downshift to Rutherford 0 or 1.
Improvement of the walking perimeter at 1 and 2 years (<200m,> 200m, unlimited) | 1 and 2 years
  Improvement of the walking perimeter is related to Rutherford stage. It is assessed by questioning the patient about the ability to have an unlimited walking distance, or moderately limited (> 200m), or severely limited (<200m).
The increase in the systolic pressure index at discharge from hospital, then at 1, 6, 12 and 24 months (<0.75,> 0.75) | 1, 6, 12 and 24 months
  The increase of the systolic pressure index (SPI) is obtained by comparing all post-operative measures to pre-operative values.
The quality of life measured by the Vascu-Qol 6 to 2 years | 2 years
  The quality of life assessment is obtained by filling the Vascu-Qol questionnaire and comparing the score with the preoperative value.
The treatment burden measured by the Treatment Burden Questionnaire at 6 months | 6 months
  The treatment burden is evaluated by comparing the Treatment Burden Questionnaire score at 6 months with the preoperative value.
Number of participants with adverse events as assessed by hematoma, redo surgery or vascular infection at 2 years | During 2 years
  Tolerance is assessed by looking for the following events during the two postoperative years: hematoma that necessitated hospital stay, vascular infection, or redo surgery because of vascular complication.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph TOUMA, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (16):
- France (16):
  - CHU - Hôpitaux de Bordeaux, Bordeaux
  - Hôpital Ambroise Paré, APHP, Boulogne-Billancourt
  - Hôpital de la Cavale Blanche, Brest
  - Centre hospitalier René Dubos, Cergy-Pontoise
  - Hôpital Henri Mondor, APHP, Créteil
  - Hôpital François Mitterrand, Dijon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Timone, APHP, Marseille
  - CHU de Nice, Nice
  - CHU Carémeau, Nîmes
  - Hôpital Européen Georges Pompidou, APHP, Paris
  - Hôpital Bichat - Claude Bernard, APHP, Paris
  - Hôpital La Pitié-Salpêtrière, APHP, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rangueil, Toulouse
  - Institut Lorrain du Cœur et des Vaisseaux Louis Mathieu, Vandœuvre-lès-Nancy